CLINICAL TRIAL: NCT01141400
Title: The Effect of Patient Cost-Sharing on Antidepressant and Adjunctive Therapy Use
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: CN138-587
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- depression & initial prescription for an antidepressant: A sample of adults with a diagnosis of depression and an initial prescription fill for an antidepressant

SUMMARY:
The primary objective of this study is to measure the effects of patient cost-sharing on the initiation of adjunctive treatment and subsequent healthcare utilization and expenditures among a population of commercially insured adults on antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18-64) will be selected from the MarketScan Commercial Database between January 1, 2004, and September 30, 2008, if they have at least two medical claims with a diagnosis of depression and at least one prescription fill for an antidepressant medication.

Exclusion Criteria:

* Patients who have any claim with a diagnosis of dementia, schizophrenia, delusional disorder, psychoses, pervasive development disorder, mental retardation, cerebral degenerations, Parkinson's disease, senility, manic depression, bipolar disorder, or major depressive disorder with psychotic symptoms.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be selected from the MarketScan Commercial Database between January 1, 2004 and September 30, 2008 (the last month of data available)
Sampling Method: Non-Probability Sample
Enrollment: 48865 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is any use of adjunctive treatment (combined and by class) and the time to initiation of adjunctive treatment (combined and by class). | 16 months
  16 months of medical and prescription drug coverage after the initial antidepressant prescription claim

SECONDARY OUTCOMES:
sensitivity to cost-sharing will be examined as a function of treatment resistance | 16 months
  16 months of medical and prescription drug coverage after the initial antidepressant prescription claim

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm